CLINICAL TRIAL: NCT03916666
Title: Chronic Low Back Pain - Epiduroscopy Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pavol Jozef Safarik University (Other)
Collaborators: Europainclinics z.ú. (Other)
Responsible Party: Principal Investigator, Kočan Ladislav, Principal investigator, Pavol Jozef Safarik University
Other Study IDs: EPCSVII
Record Dates: First submitted 2019-04-08; First posted 2019-04-16 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Epiduroscopy — Endoscopic intervention

SUMMARY:
Retrospective analysis of patients with low back pain after epiduroscopic procedure

DETAILED DESCRIPTION:
Retrospective analysis of patients with low back pain after epiduroscopic procedure Retrospective analysis of ambulatory data and next phone survey

ELIGIBILITY:
Inclusion Criteria:

* all patients after epiduroscopy

Exclusion Criteria:

* patients disagreement

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: After epiduroscopy, FBSS Y/N
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-12-11 (Estimated); Primary Completion 2021-12-11 (Estimated); Study Completion 2021-12-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of back pain after epiduroscopic procedure | 1 year
Incidence of leg pain after epiduroscopic procedure | 1 year

CONTACTS AND LOCATIONS:
Locations (2):
- EuroPainClinics .z.ú, Prague, Smetanovo Nábřeží 327/14, Czechia
- East Slovak Institute for Cardiovascular Diseases, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No